CLINICAL TRIAL: NCT07058129
Title: Deep Cervical Lymphatic Venous Anastomosis in Treatment of Alzheimer's Disease: A Multicenter, Prospective, Registry (CLEAN-AD Registry)
Brief Title: Deep Cervical Lymphatic Venous Anastomosis in the Treatment of Alzheimer's Disease (CLEAN-AD Registry)
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, yilong Wang, Professor, Beijing Tiantan Hospital
Other Study IDs: KY2025-090-02
Record Dates: First submitted 2025-05-11; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Alzheimers Disease
Keywords: Alzheimers disease; Cervical lymphatic venous anastomosis; Registry
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Deep cervical lymphatic venous anastomosis — The intervention requires to perform bilateral deep cervical lymphatic venous anastomosis (DC-LVA). Through cervical incision, the deep cervical lymphatic tissue is anatomically dissected and anastomosed with the venous system of the neck. Under indocyanine green (ICG) navigation, the flow of lymphatic fluid into the vein could be observed via ICG tracing fluorescence after surgery.
  Other Names: lymphatic venous anastomosis

SUMMARY:
This multicenter, prospective registry is to evaluate the efficacy and safety of deep cervical lymphatic venous anastomosis (DC-LVA) in reduing the clinical dementia rating-sum of boxes (CDR-SB) score of Alzheimer's Disease (AD) patients at 12 months after surgery in the real-world.

DETAILED DESCRIPTION:
Alzheimer's Disease (AD) is a common neurodegenerative disorder affecting the elderly population. Global health data estimates that there are 50 million AD patients worldwide, and this number may triple to 150 million cases by 2050. Anti-amyloid β (Aβ) monoclonal antibodies have emerged as disease-modifying therapies for preclinical or mild AD, but the majority of candidate agents have failed to demonstrate clinical efficacy. A series of case studies has suggested the efficacy of deep cervical lymphatic venous anastomosis (DC-LVA) in AD patients, however, there is currently a lack of large-sample cohort study in the real-world.

The primary purpose of this study is to evaluate the efficacy and safety of deep cervical lymphatic venous anastomosis (DC-LVA) in improve the cognitive function of AD patients at 12 months, and to identify subgroups asscociated with the treatment outcome.

This cohort is a multicenter, prospective, registry. A total of 814 patients received DC-LVA treatment in 40 centers from China will be enrolled. Face to face interviews will be made at baseline, 7 days (or hospital discharge), 3 months ± 7 days, 6months ± 15 days, 12 month ± 15 days, 18 month ± 15 days, and 24 month ±15 days.

The change of clinical dementia rating-sum of boxes (CDR-SB) score, Neuropsychiatric Inventory (NPI) score, Activities of Daily Living (ADCS-ADL) score, Caregiver Burden (ZCI-AD) score, Mini-Mental State Examination (MMSE) score, AD Assessment Scale-Cognitive Subscale (ADAS-cog13) score at 3, 6, 12, 18, 24 months, and the change of brain amyloid burden evaluated by Aβ PET-CT centiloid value at 12 months will be measured.

The changes of CDR-SB score will be analyzed using a repeated measures mixed-effects model. Least squares means will be used to estimate the levels at each time point, and the mean difference with 95% confidence intervals will be calculated. Safety outcomes will be summarized using counts/percentages. Adverse events and serious adverse events will be summarized.

In exploratory outcome measures, we will analyse the AD associated biomarkers in lymphatic tissue during the surgery, the change of fluid biomarkers (peripheral blood, saliva, urine,and cerebrospinal fluid AD associated biomarkers), the change of MRI brain volumes (total brain volume, hippocampal volume, lateral ventricle volume), the change of glymphatic function index(DTI-ALPS), the change of MRS metabolic markers (N-Acetylaspartate, Creatine, Choline, Lactate, Glutamate and Glutamine, myo-Inositol), and the change of artificial intelligence-assisted oculomotor/gait measurements during 12 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, male or famale.
2. Diagnosed with AD according to the NIA-AA criteria.
3. Patients who have received DC-LVA treatment;
4. Signed informed consent (by the subject or their relative, and caregiver)

Exclusion Criteria:

1. Severe neurological deficits in limb movement, language, vision, hearing, or consciousness, or any condition that the investigator determines may prevent the completion of cognitive function assessments.
2. The subject lacks a stable and reliable caregiver to accompany with them during entire study follow-up visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AD patients who received DC-LVA treatment
Sampling Method: Non-Probability Sample
Enrollment: 814 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2028-07-30 (Estimated); Study Completion 2029-07-30 (Estimated)

PRIMARY OUTCOMES:
The change of Clinical Dementia Rating-Sum of Boxes score at 12th months after surgery | From baseline to 12th months after surgery
  The change of Clinical Dementia Rating-Sum of Boxes score (CDR-SB, 0-18 score, higher scores mean a worse outcome)
The incidence of perioperative complications within 7 days after surgery | From baseline to 7th days after surgery
  The incidence of perioperative complications

SECONDARY OUTCOMES:
The Change of Clinical Dementia Rating-Sum of Boxes score | From baseline to 3th, 6th, 18th, 24th months after surgery
  Clinical Dementia Rating-Sum of Boxes score (CDR-SB, 0-18 score, higher scores mean a worse outcome)
The Change of Neuropsychiatric Inventory Score | From baseline to 3th, 6th, 12th,18th, 24th months after surgery
  Neuropsychiatric Inventory Score (NPI, 0-144 score, higher scores mean a worse outcome)
The Change of Alzheimer's Disease Assessment Scale-Activity of Daily Living score | From baseline to 3th, 6th, 12th, 18th, 24th months after surgery
  Alzheimer's Disease Assessment Scale-Activity of Daily Living score (ADAS-ADL, 0-78 score, higher scores mean a better outcome)
The Change of Zarit Caregiver Interview of Alzheimer's Disease Score | From baseline to 3th, 6th, 12th,18th, 24th months after surgery
  Zarit Caregiver Interview of Alzheimer's Disease Score (ZCI-AD, 0-88 score, higher scores mean a worse outcome)
The Change of Mini-Mental State Examination Score | From baseline to 3th, 6th, 12th, 18th, 24th months after surgery
  Mini-Mental State Examination Score (MMSE, 0-30 score, higher scores mean a better outcome)
The Change of Alzheimer's Disease Assessment Scale Cognitive Score | From baseline to 3th, 6th, 12th,18th, 24th months after surgery
  Alzheimer's Disease Assessment Scale Cognitive score (ADAS-Cog-13, 0-85 score, higher scores mean a worse outcome)
The Change of Aβ PET-CT Centiloid value | From baseline to 12th months after surgery
  The change of Aβ PET-CT Centiloid value at 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hopital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No